CLINICAL TRIAL: NCT02946294
Title: A Comparative Study for Evaluation of the Analgesic Profile of Ultrasound-Guided Modified Pectoral Nerves Block Versus Serratus Plane Block in Major Breast Cancer Surgery
Brief Title: Modified Pectoral Nerves Block Versus Serratus Plane Block in Major Breast Cancer Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Mostafa Kamel, Assistant Lecturer of Anesthesia and Pain Relief, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD2010014055.3; IRB00004025 (Other: Institutional Review Board)
Record Dates: First submitted 2016-10-23; First posted 2016-10-27 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- modified pectoral nerves block (Active Comparator): Modified pectoral nerves block with general anesthesia. Using the ultrasound, 10 ml of bupivacaine 0.25% with epinephrine 5 ug/ml will be injected in the plane between the pectoralis major and minor muscles. And another 20 ml of bupivacaine 0.25% with epinephrine 5 ug/ml will be injected in the plane between the pectoralis minor and the serratus anterior muscles.
  Interventions: Drug: Bupivacaine 0.25% with epinephrine
- serratus plane block (Active Comparator): Serratus plane block with general anesthesia. Using the ultrasound, 0.4 ml of bupivacaine 0.25% with epinephrine 5 ug/ml will be injected in the plane between the serratus anterior muscle and the underlying ribs.
  Interventions: Drug: Bupivacaine 0.25% with epinephrine

INTERVENTIONS:
Drug: Bupivacaine 0.25% with epinephrine
  Other Names: Markyrene
  Arms: modified pectoral nerves block
Drug: Bupivacaine 0.25% with epinephrine
  Other Names: Markyrene
  Arms: serratus plane block

SUMMARY:
The purpose of this study is to compare the analgesic profile of modified pectoral nerves block and serratus plane block in patients undergoing mastectomy.

DETAILED DESCRIPTION:
This study includes three groups. The first group will receive ultrasound-guided modified pectoral nerves block prior to induction of general anesthesia. The second one will receive ultrasound-guided serratus plane block prior to induction of general anesthesia. The third one will not receive any block preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists( ASA) I or II and scheduled for major breast cancer surgery( modified radical mastectomy or conservative mastectomy with axillary evacuation).

Exclusion Criteria:

* Local infection at the site of the block, coagulations abnormalities, allergy to local anesthetics or morphine, body mass index> 35, patient refusal, severe respiratory or cardiac disorders, pre-existing neurological deficits, hepatic or renal insufficiency, chronic pain syndrome, chronic analgesic use and psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption | Intraoperative
Total morphine consumption | The first 24 hours postoperative
Visual analogue scale score at rest and during shoulder movement | The first 24 hours postoperative

SECONDARY OUTCOMES:
Mean arterial blood pressure | Preincision, 1 minute postincision, 1 hour postincision, 4, 8, 12, 24 hours postoperative
  Hemodynamics
Heart rate | Preincision, 1 minute postincision, 1 hour postincision, 4, 8, 12, 24 hours postoperative
  Hemodynamics
Time to first requirement of rescue analgesia | The first 24 hours postoperative
Sedation score | Immediate postoperative, 1, 4, 8, 12, 24 hours postoperative
  as a side effect of morphine
Respiratory rate | Immediate postoperative, 1, 4, 8, 12, 24 hours postoperative
  respiratory depression defined as respiratory rate <12 breaths per minute
Nausea and vomiting | The first 24 hours postoperative
  as a side effect of morphine
Patient satisfaction with postoperative analgesia | One week after surgery
  using numerical rating scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Ghoneim, MD, Study Director — National Cancer Institute, Cairo University; Ahmad H Aboul Soud, MD, Study Chair — National Cancer Institute, Cairo University; Khaled M Salem, Master, Principal Investigator — National Cancer Institute, Cairo University; Mohamed E Hassan, MD, Principal Investigator — National Cancer Institute, Cairo University; Ahmad H Mohamed, MD, Principal Investigator — National Cancer Institute, Cairo University
Locations (1):
- National Cancer Institute, Cairo, Misr Al Qadimah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hards M, Harada A, Neville I, Harwell S, Babar M, Ravalia A, Davies G. The effect of serratus plane block performed under direct vision on postoperative pain in breast surgery. J Clin Anesth. 2016 Nov;34:427-31. doi: 10.1016/j.jclinane.2016.05.029. Epub 2016 Jun 16. PMID 27687427
- [Background] Zocca JA, Chen GH, Puttanniah VG, Hung JC, Gulati A. Ultrasound-Guided Serratus Plane Block for Treatment of Postmastectomy Pain Syndromes in Breast Cancer Patients: A Case Series. Pain Pract. 2017 Jan;17(1):141-146. doi: 10.1111/papr.12482. Epub 2016 Sep 2. PMID 27587333
- [Background] Mayes J, Davison E, Panahi P, Patten D, Eljelani F, Womack J, Varma M. An anatomical evaluation of the serratus anterior plane block. Anaesthesia. 2016 Sep;71(9):1064-9. doi: 10.1111/anae.13549. Epub 2016 Jul 20. PMID 27440171
- [Background] Okmen K, Okmen BM, Uysal S. Serratus Anterior Plane (SAP) Block Used for Thoracotomy Analgesia: A Case Report. Korean J Pain. 2016 Jul;29(3):189-92. doi: 10.3344/kjp.2016.29.3.189. Epub 2016 Jul 1. PMID 27413485
- [Background] Daga V, Narayanan MK, Dedhia JD, Gaur P, Crick H, Gaur A. Cadaveric feasibility study on the use of ultrasound contrast to assess spread of injectate in the serratus anterior muscle plane. Saudi J Anaesth. 2016 Apr-Jun;10(2):198-201. doi: 10.4103/1658-354X.168825. PMID 27051373
- [Background] Khemka R, Chakraborty A, Ahmed R, Datta T, Agarwal S. Ultrasound-Guided Serratus Anterior Plane Block in Breast Reconstruction Surgery. A A Case Rep. 2016 May 1;6(9):280-2. doi: 10.1213/XAA.0000000000000297. PMID 26934607
- [Background] Bhoi D, Pushparajan HK, Talawar P, Kumar A, Baidya DK. Serratus anterior plane block for breast surgery in a morbidly obese patient. J Clin Anesth. 2016 Sep;33:500-1. doi: 10.1016/j.jclinane.2015.09.004. Epub 2015 Oct 23. No abstract available. PMID 26603109
- [Background] Ohgoshi Y, Yokozuka M, Terajima K. [Serratus-Intercostal Plane Block for Brest Surgery]. Masui. 2015 Jun;64(6):610-4. Japanese. PMID 26437549
- [Background] Madabushi R, Tewari S, Gautam SK, Agarwal A, Agarwal A. Serratus anterior plane block: a new analgesic technique for post-thoracotomy pain. Pain Physician. 2015 May-Jun;18(3):E421-4. PMID 26000690
- [Background] Kunhabdulla NP, Agarwal A, Gaur A, Gautam SK, Gupta R, Agarwal A. Serratus anterior plane block for multiple rib fractures. Pain Physician. 2014 Sep-Oct;17(5):E651-3. No abstract available. PMID 25247916
- [Background] Eid M. Other potential uses of serratus anterior plane block. Anaesthesia. 2014 Aug;69(8):933-4. doi: 10.1111/anae.12778. No abstract available. PMID 25039953
- [Background] Kikuchi M, Takaki S, Nomura T, Goto T. [Difference in the Spread of Injectate between Ultrasound Guided Pectoral Nerve Block I and II. A Cadaver Study]. Masui. 2016 Mar;65(3):314-7. Japanese. PMID 27097516
- [Background] Tan YR, Quek KH. Tackling the axillary blind spot with PECS II. Anaesthesia. 2015 Feb;70(2):230-1. doi: 10.1111/anae.13005. No abstract available. PMID 25583191
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Purcell N, Wu D. Novel use of the PECS II block for upper limb fistula surgery. Anaesthesia. 2014 Nov;69(11):1294. doi: 10.1111/anae.12876. No abstract available. PMID 25302976
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Derived] Bakeer AH, Kamel KM, Abdelgalil AS, Ghoneim AA, Abouel Soud AH, Hassan ME. Modified Pectoral Nerve Block versus Serratus Block for Analgesia Following Modified Radical Mastectomy: A Randomized Controlled Trial. J Pain Res. 2020 Jul 14;13:1769-1775. doi: 10.2147/JPR.S252539. eCollection 2020. PMID 32765052